CLINICAL TRIAL: NCT05263154
Title: Goal-directed Low vs. High Oxygen Therapy During Anesthesia for Abdominal Surgery
Brief Title: Goal-directed Low Oxygen During Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Karl A Franklin, Profesor, Consultant surgeon, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-02211
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Complications
Keywords: postoperative hypoxia; abdominal surgery; randomized controlled trial
MeSH Terms: conditions — Postoperative Complications | interventions — high-potential iron-sulfur protein oxygen oxidoreductase

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal directed low oxygen (Experimental): Oxygen given at low concentrations following goals of oxygen saturation during and after anesthesia
  Interventions: Other: Goal directed low oxygen
- High oxygen (Active Comparator): Oxygen given as traditionally including high concentrations
  Interventions: Other: High oxygen

INTERVENTIONS:
Other: Goal directed low oxygen — Oxygen is titrated until oxygen saturation is 100% in one-minute steps before the induction of anesthesia, with increasing fraction of inspired oxygen (FiO2) from 0.25 to 0.30 to 0.35 and so on. After intubation, the FiO2 is set to 0.25 to achieve a target saturation of 94-96%. Supplementary oxygen after surgery will be given with the same targets and with as little oxygen as necessary.
  Arms: Goal directed low oxygen
Other: High oxygen — FiO2 1.0 before induction until end-tidal oxygen concentrations of 0.80 occur. The FiO2 will be reduced to 0.35 during anesthesia, followed by an increase in FiO2 to 0.80 during 5 minutes before extubating the patient, followed by FiO2 0.40 for at least thirty minutes after anesthesia. Oxgen will then be given at 3 liters a minute with a oxygen saturation goal of 98%
  Arms: High oxygen

SUMMARY:
The study aims at investigate whether low oxygen therapy during anesthesia improves oxygen partial pressure and lung function in the postoperative period after abdominal surgery. 200 patients scheduled for abdominal surgery will be randomized (1:1) to goal directed low oxygen concentration during and after anesthesia vs. fixed high oxygen concentration. Arterial oxygen partial pressure is the primary outcome and lung function a secondary explanatory outcome.

DETAILED DESCRIPTION:
Postoperative hypoxia is a most common complication after major abdominal surgery. This study aims at investigate whether goal-directed low oxygen therapy during anesthesia improves oxygen partial pressure and lung function in the postoperative period after abdominal surgery.

200 adult patients scheduled for major abdominal cancer surgery lasting for more than 2 hours will be included after signed informed consent. Patients will then be randomized to either goal directed low oxygen or high oxygen during anesthesia and in the postoperative period.

Patients who are randomized to goal directed low oxygen will be given oxygen before the induction of anesthesia, with increasing fraction of inspired oxygen (FiO2) from 0.25 to 0.30 to 0.35 and so on. After intubation, the FiO2 is set to 0.25 to achieve a target saturation of 94-96%. Supplementary oxygen after surgery will be given with the same targets and with as little oxygen as necessary, Patients who are randomized to high oxygen will be given FiO2 of 1.0 before induction until end-tidal oxygen concentrations of 0.80 occur. The FiO2 will be reduced to 0.35 during anesthesia, followed by an increase in FiO2 to 0.80 during 5 minutes before extubating the patient, followed by FiO2 0.40 for at least thirty minutes after anesthesia. Oxgen will then be given at 3 liters a minute with a oxygen saturation goal of 98%.

Arterial blood gases, lung function measurements including diffusion capacity will be taken on the day before surgery. Blood gases will be taken during the first and second day after surgery and lung function tests during the second day after surgery. Blood gases and lung function will also be obtained at three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being scheduled for a major abdominal cancer surgery lasting for more than 2 hours.
* Having a condition within American Society of Anesthesia Class 1-3.

Exclusion Criteria:

* Being at risk for a difficult intubation during anesthesia in the form of Mallampati score 3-4, or having a previous documentation of difficult intubation.
* Decline participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in arterial oxygen partial pressure after surgery vs. before surgery | 3 days
  Oxygen partial pressure

SECONDARY OUTCOMES:
Mean change in diffusion capacity for carbon-monoxide after surgery vs. before surgery | 3 days
  Diffusion capacity
Mean change in vital capacity after surgery vs. before surgery | 3 days
  Vital capacity
Mean change in forced expiratory volume in one second after surgery vs. before surgery | 3 days
  Forced expiratory volume in one second
Mean change in arterial carbon-dioxide partial pressure after surgery vs. before surgery | 3 days
  Carbon-dioxide partial pressure
Mean change in arterial oxygen partial pressure after surgery vs. before surgery | 3 months
  Oxygen partial pressure
Mean change in diffusion capacity for carbon-monoxide after surgery vs. before surgery | 3 months
  Diffusion capacity
Mean change in vital capacity after surgery vs. before surgery | 3 months
  Vital capacity
Mean change in forced expiratory volume in one second after surgery vs. before surgery | 3 months
  Forced expiratory volume in one second
Mean change in arterial carbon-dioxide partial pressure after surgery vs. before surgery | 3 months
  Carbon-dioxide partial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- University hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No
Depends on what is allowed according to Swedish Ethical authority.